CLINICAL TRIAL: NCT01313507
Title: Clinical Study to Evaluate the Safety and Tolerability of Immunoglobulin Intravenous (Human) 10% (NewGam) Administered at High Infusion Rates to Patients With Primary Immunodeficiency Diseases (Extension of Study NGAM-01)
Brief Title: High Infusion Rate Study of Immunoglobulin Intravenous (Human) 10% (NewGam)
Acronym: NGAM-05
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGAM-05
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Primary Immunodeficiency Disease
Keywords: Primary Immunodeficiency Disease; PID
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NewGam (Experimental): Participants received NewGam 200-800 mg/kg intravenously every 3 or 4 weeks for 3 months (5 or 4 total infusions, respectively).
  Interventions: Biological: NewGam

INTERVENTIONS:
Biological: NewGam — The initial dose and dosing interval for each participant was the dose and dosing interval the participant received at the end of the NGAM-01 study. The dose of NewGam, solvent/detergent treated human normal immunoglobulin 10%, remained the same throughout the study, as long as the minimum trough level of serum immunoglobulin G (IgG) was above 5 g/L. If the serum IgG trough level dropped to 5 g/L or less, the dose was to be adjusted at the investigator's discretion. NewGam was supplied as a solution for infusion.

SUMMARY:
This was a prospective, open-label, non-controlled, non-randomized multicenter Phase III study of 2 multiple-dose intravenous NewGam regimens (every 3 weeks or every 4 weeks, continuing the patient's infusion interval in the main study NCT01012323 [NGAM-01]) for 3 months. The primary objective of the study was to assess the safety and tolerability of high infusion rates of NewGam.

DETAILED DESCRIPTION:
Patients received NewGam via an infusion pump to control precise infusion rates. All NewGam infusions started at a rate of 0.01 mL/kg/min (60 mg/kg/h) for the first 30 minutes followed by 0.03 mL/kg/min (180 mg/kg/h) for the next 15 minutes. If tolerated, further increments were made at predefined patterns with the following maximum rates: 0.10 mL/kg/min (600 mg/kg/h) in the first infusion; if this was tolerated, 0.12 mL/kg/min (720 mg/kg/h) in the second infusion; if this was tolerated, 0.14 mL/kg/min (840 mg/kg/h) in all subsequent infusions.

If an adverse event occurred during an infusion, the rate was reduced to half the rate at which the event occurred or the infusion was interrupted until symptoms subsided. The infusion was then resumed at a rate tolerated by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the main study NGAM-01.
* At each of the last 3 infusions in the main study NGAM-01, administration of NewGam at the maximum infusion rate of 0.08 mL/kg/min and without the need for premedication.

Exclusion Criteria:

* Any condition or circumstance that would have led to the exclusion of the subject from the NGAM-01 study.
* Administration of any immunoglobulin infusion other than NewGam between conclusion of the NGAM-01 study and the beginning of the present study.
* A deviation of the subject's treatment interval of more than 7 days between the last infusion of NewGam in the NGAM-01 study and the first infusion of NewGam in the present study.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James N Moy, MD, Principal Investigator — Rush Medical Center
Locations (6):
- United States (6):
  - University of California Irvine, Irvine, California
  - Immunoe Research Center, Centennial, Colorado
  - Rush Universtity Medical Center, Chicago, Illinois
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Midlands Pediatrics, Papillion, Nebraska
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NewGam
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: All participants who received at least 1 dose of NewGam.
Arm/Group | NewGam
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.8 (19.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in the Quality of Life (QoL) at the End of the Study
Description: QoL was assessed with the Child Health Questionnaire-Parent Form (CHQ-PF50), completed by a parent or guardian, in participants < 14 years of age at the start of the previous study NGAM-01 and with the Short Form-36 Health Survey (SF-36-HS) in participants ≥ 14 years of age. The CHQ-PF50 consists of 50 items organized into 15 subscales.The 15 subscales could be combined into 2 summary scores, physical and psychosocial. The calculated scores were transformed so that each scale had a range of 0-100. A higher score indicates better health. The SF-36-HS is composed of 36 items. Responses to the 36 items were combined to create 8 scales. The 8 scales could be further combined into 2 scores: Physical component summary and mental component summary. The item and scale scores were transformed to a range of 0-100 with a mean of 50 and a standard deviation of 10 in the general US population. A higher score indicates better health. For both instruments, a positive change indicates improvement.
Time Frame: Baseline (follow-up visit of study NGAM-01) to the end of the study (follow-up visit of study NGAM-05) (up to 4 months)
Population: Safety analysis set: All participants who received at least 1 dose of NewGam.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | NewGam
Number analyzed (Participants) | 21
Units on a scale
  CHQ-PF50 - Physical component summary | -2.63 (5.22)
  CHQ-PF50 - Psychosocial component summary | -2.01 (5.78)
  SF-36 - Physical component summary | 0.21 (6.00)
  SF-36 - Mental component summary | 0.36 (7.33)

2. Primary Outcome: Percentage of Participants Who Experienced at Least 1 Adverse Event Causally Related to the Administration of the Study Drug
Description: An adverse event was considered to be causally related to the administration of the study drug if it judged to be probably or possibly related to the study drug, as assessed by the investigator.
Time Frame: Baseline (follow-up visit of study NGAM-01) to the end of the study (follow-up visit of study NGAM-05) (up to 4 months)
Population: Safety analysis set: All participants who received at least 1 dose of NewGam.
Measure: Number; unit: Percentage of participants
Arm/Group | NewGam
Number analyzed (Participants) | 21
Percentage of participants | 19.0

3. Primary Outcome: Percentage of Participants Who Experienced at Least 1 Adverse Event Temporally Related to the Study Drug
Description: An adverse event was considered to be temporally related to the study drug if it started during an infusion or within 72 hours after the end of an infusion.
Time Frame: Baseline (follow-up visit of study NGAM-01) to the end of the study (follow-up visit of study NGAM-05) (up to 4 months)
Population: Safety analysis set: All participants who received at least 1 dose of NewGam.
Measure: Number; unit: Percentage of participants
Arm/Group | NewGam
Number analyzed (Participants) | 21
Percentage of participants | 38.1

ADVERSE EVENTS:
Description: Safety analysis set: All participants who received at least 1 dose of NewGam.
Arm/Group | NewGam
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 12/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NewGam (N=21)
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Chest pain (General disorders) | 2
Pyrexia (General disorders) | 2
Sinusitis (Infections and infestations) | 4
Headache (Nervous system disorders) | 2
Nasopharyngitis (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Octapharma agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Octapharma supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial. Octapharma also reserves the right to review data prior to publishing and provide comments/changes within a certain time period.